CLINICAL TRIAL: NCT05576987
Title: The Effect of the Health Belief Model-Based Intervention in Primary School 3rd and 4th Grade Students' Behavior on Safety Precautions for Preventing Accidents at School
Brief Title: Student Behavior in School Accident Precautions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Afyonkarahisar Health Sciences University (Other)
Responsible Party: Principal Investigator, Cahide Çevik, Assistant professor, Afyonkarahisar Health Sciences University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: İnterventional
Record Dates: First submitted 2022-09-26; First posted 2022-10-13 (Actual); Results first posted 2026-01-08 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-12

CONDITIONS: Health Behavior
Keywords: schools; accident; students; health belief model
MeSH Terms: conditions — Health Behavior | interventions — Educational Status

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Experimental): Experimental group will be selected from the branches 3rd and 4th grade. 3 branches will be selected for the experimental group. Branches will be determined by drawing. In order not to interfere with the education of students during the training, the groups will be designated as class branches.
  Interventions: Behavioral: Education
- control group (No Intervention): Control group will be selected from the branches 3rd and 4th grade. 3 branches for the control group. Branches will be determined by drawing. In order not to interfere with the education of students during the training, the groups will be designated as class branches.
  After the training of the experimental group is completed and the final data are obtained, a 40-minute training will be given to the control group about prevention from school accidents. This training was planned so that the control group would not be devoided of the intervention.

INTERVENTIONS:
Behavioral: Education — Students selected for the experimental group will be trained by the researcher for school accidents prepared in line with the components of the Health Belief Model.The training program will be planned as 30 minutes per week for 4 weeks. Before the training and at the end of the training (at the end of the 4th week), the students will be applied personal information form and a behavior scale for safety precautions in school accidents.
  Arms: intervention group

SUMMARY:
Accidents are an important public health problem due to temporary or permanent disability and deaths. Injuries are among the most important causes of death and lifelong disability between the ages of 5-14. Children at these ages spend long hours at school and are physically very active in school. It is reported that 15% of child accidents occur at school. For this reason, it is important to increase the standard of knowledge of children to improve their behavior towards safety precautions.

Purpose of this study is to research the impact of the education that has given towards the health belief model, for the behavior of children about precautions against school accidents. This study is Quasi-experimental study. There will a experiment and a control group in the study. Within the scope of the study, the researcher will train students about school accidents and how to prevent them for 30 minutes a week at the total of 4 weeks. No intervention will be applied to the control group. The scale will be applied to the students, before the training and afterwards to determine the behaviors of students towards safety precautions in school accidents.

DETAILED DESCRIPTION:
The behavior score averages and standard deviations of the two groups in a previous study (Dilek, 2018) and the effect size were calculated to determine the sample size of the study. Power analysis (significance level 0.05 for type 1 error, effect size 0.50, and power 0.95). (Gpower 3.1 version) was carried out. In the power analysis, the minimum number of participants was 87 in the experimental group and 87 in the control group.

In this context, the research will be conducted with 100 participants in each group, taking into account the possibility that non-parametric statistics may need to be used due to the non-normal distribution of the dependent variable, incomplete and erroneous data, and absenteeism.

Experimental and control groups will be selected from the branches 3rd and 4th grade. 3 branches will be selected for the experimental group and 3 branches for the control group. Branches will be determined by drawing. In order not to interfere with the education of students during the training, the groups will be designated as class branches.

Ethical permission was obtained from the Ethics Committee of Afyonkarahisar Sağlık Bilimleri Üniversitesi (Afyonkarahisar Health Sciences University) (date: 03.June 2022; Number: 2022/340)

ELIGIBILITY:
Inclusion Criteria:

* Being educated in 3rd and 4th grade
* Volunteer to participate in the research
* Consent of the student's parent
* Speak and understand Turkish

Exclusion Criteria:

* Being visually and hearing impaired
* Using a language other than Turkish
* Not willing to participate in the study

Ages: 9 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 200 (Actual)
Dates: Start 2022-10-05 (Actual); Primary Completion 2022-10-26 (Actual); Study Completion 2022-10-26 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Afyonkarahisar Health Sciences University, Afyonkarahisar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Study using data for power analysis — https://acikbilim.yok.gov.tr/bitstream/handle/20.500.12812/30971/yokAcikBilim_10181723.pdf?sequence=-1&isAllowed=y
- See also: The research that conducted the validity and reliability study of the scale used in the study — https://tez.yok.gov.tr/UlusalTezMerkezi/tezSorguSonucYeni.jsp

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was carried out in a primary school. The study began with 100 students in each group. 3 branches were selected for the experimental group and 3 branches for the control group. Branches were determined by lottery. The students to be included in the experimental group were selected from 3 branches. The students to be included in the control group were also selected from the other 3 branches.
Units Other Than Participants: School Branches
Period: Overall Study
Arm/Group | Intervention Group | Control Group
Started | 100; 3 School Branches (At the beginning of the study, a personal data form and a behavioral scale for safety measures in school accidents were applied to the students selected in the experimental group. Afterwards, the training prepared for school accidents in line with the components of the Health Belief Model (SIM) was given by the researcher for 20 minutes once a week for 4 weeks.) | 100; 3 School Branches (At the beginning of the study, a personal data form and a behavioral scale for safety measures in school accidents were applied to the students selected for the control group. No other intervention was made.)
Completed | 90; 3 School Branches (After the educational intervention was completed (4 weeks later), the personal data form and the behavior scale for safety measures in school accidents were applied again. Due to various reasons, 10 students did not attend some of the educational sessions. The data of the students who participated in four training sessions were analyzed.) | 92; 3 School Branches (After 4 weeks, the personal data form and the behavior scale for safety measures in school accidents were applied again. After the data were obtained at the end of the study, the students in the control group were also given education about school accidents (so that they would not be deprived of the training given to the experimental group). Eight students refused to respond to the scale for the post-test data.)
Not Completed | 10; 0 School Branches | 8; 0 School Branches

BASELINE CHARACTERISTICS:
Population: Due to absenteeism during various weeks of the training sessions, 10 students who did not complete the training were excluded from the study. Data from 90 students who attended all sessions over four consecutive weeks were included in the analysis. In the control group, 8 students did not complete the second assessment following the initial scale administration and were therefore excluded. The study was completed with 92 participants in the control group.
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention Group | Control Group | Total
Number analyzed (Participants) | 90 | 92 | 182
Age, Categorical [Count of Participants; unit: Participants] — Population: 10 students in the intervention Group group and 7 students in the control group left the study voluntarily. For this reason, data of 90 students in the intervention Groupgroup and 92 students in the control group were analyzed.
  Participants
    <=18 years | 90 | 92 | 182
    Between 18 and 65 years | 0 | 0 | 0
    >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Due to absenteeism during various weeks of the training sessions, 10 students who did not complete the training were excluded from the study. Data from 90 students who attended all sessions over four consecutive weeks were included in the analysis. In the control group, 8 students did not complete the second assessment following the initial scale administration and were therefore excluded. The study was completed with 92 participants in the control group
  years | 9.4 (0.64) | 9.2 (0.79) | 9.3 (0.72)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Due to absenteeism during various weeks of the training sessions, 10 students who did not complete the training were excluded from the study. Data from 90 students who attended all sessions over four consecutive weeks were included in the analysis. In the control group, 8 students did not complete the second assessment following the initial scale administration and were therefore excluded. The study was completed with 92 participants in the control group
  Participants
    Female | 41 | 44 | 85
    Male | 49 | 48 | 97
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: Participants] — Population: Due to absenteeism during various weeks of the training sessions, 10 students who did not complete the training were excluded from the study. Data from 90 students who attended all sessions over four consecutive weeks were included in the analysis. In the control group, 8 students did not complete the second assessment following the initial scale administration and were therefore excluded. The study was completed with 92 participants in the control group
  Participants
    Turkey | 90 | 92 | 182

OUTCOME MEASURES:

1. Primary Outcome: Behavior Towards The Security Precautions Against School Accidents
Description: Students' behaviors regarding safety measures in school accidents were measured through a scale. A total score was obtained based on students' responses to the scale. Statistical analysis was conducted according to the obtained scores.
  The information related to the scale is provided below. Scale of Behavior Towards The Security Precautions Against School Accidents: Student behaviors will be determined with this scale. It is a 5-point Likert-type scale consisting of 40 items and was developed by Gür and Yıldız (2009). The scale allows for a minimum score of 40 and a maximum score of 200. The highest score obtained from the scale indicates that the student has taken safety measures for school accidents at the highest level.
Time Frame: The scale was applied once at the beginning of the study and again at the end of the study (4th week).
Measure: Mean (Standard Deviation); unit: Scale score
Groups:
- Control Group: Control group will be selected from the branches 3rd and 4th grade. 3 branches for the control group. Branches will be determined by drawing. In order not to interfere with the education of students during the training, the groups will be designated as class branches.
  The students in these branches will constitute the study sample.
  After the training of the experimental group is completed and the final data are obtained, a 40-minute training will be given to the control group about prevention from school accidents. This training was planned so that the control group would not be devoided of the intervention.
- Intervention Group: Experimental group will be selected from the branches 3rd and 4th grade. 3 branches will be selected for the experimental group. Branches will be determined by drawing. In order not to interfere with the education of students during the training, the groups will be designated as class branches.
  The students in these branches will constitute the study sample.
  Education: Students selected for the experimental group will be trained by the researcher for school accidents prepared in line with the components of the Health Belief Model.The training program will be planned as 30 minutes per week for 4 weeks. Before the training and at the end of the training (at the end of the 4th week), the students will be applied personal information form and a behavior scale for safety precautions in school accidents.
Arm/Group | Control Group | Intervention Group
Number analyzed (Participants) | 92 | 90
Scale score
  pretest | 134.46 (15.70) | 131.66 (17.50)
  posttest | 136.68 (17.05) | 132.73 (18.97)

ADVERSE EVENTS:
Time Frame: Adverse Events were not monitored.
Description: Adverse Events were not monitored.
Arm/Group | Intervention Group | Control Group
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-06-03): https://cdn.clinicaltrials.gov/large-docs/87/NCT05576987/Prot_SAP_000.pdf
  • Informed Consent Form (2022-06-03): https://cdn.clinicaltrials.gov/large-docs/87/NCT05576987/ICF_001.pdf